CLINICAL TRIAL: NCT06461000
Title: EULAR Impact of Rheumatic and Musculoskeletal Diseases Survey
Acronym: ImpactSurvey
Status: Recruiting | Type: Observational
Sponsor: European Alliance of Associations in Rheumatology (Other)
Responsible Party: Sponsor
Other Study IDs: EPI001
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Rheumatologic Disease; Musculoskeletal Diseases
MeSH Terms: conditions — Collagen Diseases; Musculoskeletal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survey: Usual survey
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — online survey for participants

SUMMARY:
The EULAR Impact of RMDs Survey collects first-hand information about the impact of rheumatic and musculoskeletal diseases (RMDs) among patients across and beyond Europe. Through periodic questionnaires, patients will provide information about their healthcare situation, and how the disease affects their social and occupational lives. This data will be an important resource for researchers, healthcare professionals, and patients alike, providing valuable insights into the burden of disease and helping improve the overall care for people living with these conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18-year-old at time of baseline survey
* Living in a EULAR country at time of baseline survey
* Diagnosed with at least one RMD
* Valid personal e-mail address
* Being able to use an internet website

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - adults with at least 1 RMD
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-06-12 (Estimated); Study Completion 2029-06-12 (Estimated)

PRIMARY OUTCOMES:
General population description - country | every 6 months for up to 5 years
  country of residence
General population description - diagnosis | every 6 months for up to 5 years
  diagnosis (name of the disease)
General population description | every 6 months for up to 5 years
  year of birth

SECONDARY OUTCOMES:
Diagnosis history - physician treating the RMD | every 6 months for up to 5 years
  Primary physician specialty treating the patient
Diagnosis history - outpatient care history | every 6 months for up to 5 years
  number of medical appointments for the past 6 months
Diagnosis history - timeline | every 6 months for up to 5 years
  waiting time for medical appointments and time spent in medical appointments
Diagnosis history - Inpatient care | every 6 months for up to 5 years
  number of days of hospitalization during the past 6 months.
Non-pharmacological and pharmacological treatments. | every 6 months for up to 5 years
  Names of medications taken by the patients (from a list)
Other chronic diseases | every 6 months for up to 5 years
  diagnosis of chronic diseases other than RMD and medication taken for these conditions.
Disease burden - impact of disease | every 6 months for up to 5 years
  Rheumatic Arthritis Impact of Disease (RAID) version 7 questionnaire. The RAID is calculated based on 7 Numerical rating scales (NRS) questions. Each NRS is assessed as a number between 0 and 10. The 7 NRS correspond to pain, function, fatigue, sleep, emotional well-being, physical well-being, and coping/self-efficacy. The range of the final RAID value is 0-10 where higher figures indicate worse status.
Disease burden - health assessment | every 6 months for up to 5 years
  Health assessment questionnaire version 2 (HAQ2). The HAQ comprises of 20 questions covering 20 daily activities. These are divided in eight domains: dressing and grooming, rising, eating, walking, hygiene, reaching, gripping, and other activities. Each question is scored according to a four-point scale (0-3), and the highest scores from each domain are summed and divided by eight, to derive a total HAQ score, which ranges from 0 to 3 (3 = highest level of disability).
Disease burden - quality of life | every 6 months for up to 5 years
  patient health questionnaire (PHQ-8). The PHQ-8 is a self-reported measure of depressive symptoms composed of 8 Likert type items with a response scale ranging from 0 (Not at all) to 3 (Nearly every day), that refer to the presence of that symptom during the previous 2 weeks.Each item corresponds to the first 8 symptoms of the 4th edition of the DSM-IV diagnostic criteria for major depressive disorder. The PHQ-8 final score is obtained by adding the score for each of the items, ranging from 0 to 24 (higher scores corresponding to higher levels of depression).
Consequences on work and life (WPAI questionnaire) | every 6 months for up to 5 years
  work productivity and activity impairment questionnaire (WPAI), including total number of sick leave days due to RMD in the past 6 months. Final score is calculated in % higher scores on the WPAI indicate worse outcomes
Other barriers due to RMD | every 6 months for up to 5 years
  impact on family, leisure, social and work activities (quality of life questionnaire)
Health care | every 6 months for up to 5 years
  support from professionals (general questionnaire), satisfaction with care (scale, 1= low, 5 = high satisfaction)
Demographics - persons living with patient | every 6 months for up to 5 years
  number of persons living in household
Demographics - professional status | every 6 months for up to 5 years
  professional status

CONTACTS AND LOCATIONS:
Locations (1):
- EULAR, Kilchberg, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: EULAR Impact of RMDs Survey — https://www.eular.org/eular-impact-of-rmds-survey